CLINICAL TRIAL: NCT05768789
Title: The Impact of Buoy on Hydration Status of Active Men and Women
Brief Title: Buoy Electrolyte Study on Hydration Status of Active Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Harikesh Subramanian, Assistant Professor of Anesthesiology and Perioperative Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22090018
Record Dates: First submitted 2022-10-25; First posted 2023-03-14 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Dehydration; Electrolyte Imbalance; Electrolyte Depletion; Fluid and Electrolyte Imbalance
Keywords: dehydration; electrolyte; electrolyte supplement; electrolyte loss; electrolyte ingestion; hydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: All participants received the interventions in the same order one after the other on different days (Buoy, then Water, then Nuun) to complete the 3 arms of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Buoy Electrolyte then Water only then Nuun Electrolyte (Experimental): Visit 1: Buoy intervention amount is 4% of total body weight given in 16 divided doses over 4 hours. The goal is to give 600mg of Na+ over 4 hours while measuring urine output over 6 hours. Therefore, to safely achieve a total dose 600mg Na+ (6-fold increase from single dose) we will use 4 tsps (18 ml) of Buoy diluted in 1 L of water.
  Visit 2: Water serves as a control. Participants will ingest the same quantity of water (1 L) at a rate of 6.25% of the calculated amount of water every 15 min for 4 hours.
  Visit 3: Nuun intervention given as 1L bolus and then free water in divided doses for a total of 4% total body weight. The goal is to give a one-time dose of Nuun (600mg Na+) at the start of the trial, diluted in 1L water to be consumed within 30 min (similar to prior published data, Pence 2020).
  Interventions: Dietary Supplement: Buoy Electrolyte; Other: Water only; Dietary Supplement: Nuun Electrolyte

INTERVENTIONS:
Dietary Supplement: Buoy Electrolyte — Each subject consumed Beverage 1 (Buoy Hydration Drops) at a dose containing 600 mg/L of Na+ over 4 hours while measuring urine output over 6 hours.
Other: Water only — Each subjected ingested 1 L of Kirkland® bottled water at a rate of 6.25% of the total amount of water every 15 minutes for four hours
Dietary Supplement: Nuun Electrolyte — Each subject consumed 1 L of water with two dissolved Nuun® Sport Hydration tabs (Nuun, Seattle, WA), containing 600 mg of sodium, over 30 minutes (2 equal volumes every 15 minutes) while measuring urine output over 6 hours (

SUMMARY:
Buoy is an all-natural, organic, FDA compliant dietary electrolyte supplement that can be dissolved in 8-12oz water (or other liquid) and provide electrolytes in servings of 1/3 teaspoon. This study will evaluate Buoy in hydrating active adults.

DETAILED DESCRIPTION:
Prior to initiation of the study, participants will have a screening visit to complete informed consent and health history. The history for females will include their last date for menstruation and/or birth control method to take into consideration the effects of ovulation on water retention. During this visit we will measure heart rate, blood pressure, height, weight. Females will be administered a urine pregnancy test.

Participants must refrain from vigorous exercise within 24 hours of study visit. Participants will fast (food) overnight for 10h prior to initiation of test. Upon waking they are asked to empty their bowel & bladder. They can consume one 8oz cup of coffee or other liquid. They will present at 7-8am at which time they will be asked to empty their bladder again. After resting for 5 minutes baseline vitals will be taken, including blood pressure, heart rate, weight, bioimpedance. Urinalysis dipstick for protein/blood/glucose and i-STAT measurement for creatinine and electrolytes on Visit 1 to confirm eligibility. For Visit 2 and Visit 3, the participant will be asked to review medical history and any change in status may warrant an additional baseline creatinine and blood/protein test to confirm eligibility. Additional food or beverage will not be allowed throughout the study period. All studies will be repeated in the same subject using either Buoy (intervention) or water (control) or Nuun (intervention). Urine will be collected at four specific timepoints during the intervention and the volume will be recorded. If participants need to urinate between scheduled collection times, urine will be collected, volume recorded, and combined with the urine collection of the following timepoint. These urine samples will be measured and a fraction of it will be sent to the lab to be tested for the following electrolytes: sodium, potassium, chloride and urine osmolarity. Urine creatinine will also be tested at these timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 to 45 years of age
* Freely given written consent
* Non-tobacco users
* Negative pregnancy test in women of childbearing potential
* BMI < 35 kg/m2
* GFR > 60 ml/min
* No known underlying medical condition
* Willing to refrain from EtOH for 24h prior to test day
* Willing to refrain from strenuous exercise for 24 h prior to each test day
* Acceptable to have one 8oz cup of coffee/liquid on the morning of the test, but must be consistent each visit
* Without active infection of any kind
* Engaged in exercise three or more hours per week

Exclusion Criteria:

* Abnormal creatinine (Cr > 1.2).
* Proteinuria / hematuria / glucosuria based on urine dipstick.
* Diagnosed medical condition that would impede results (CHF, HTN, CAD, CKD, history of electrolyte abnormality).
* Pregnancy
* Use of diuretics within past 2 weeks
* Obesity (BMI > 35)
* Active infection based on symptoms (bacterial or viral)
* Hemodynamic abnormality at screening visit: Blood pressure less than 100/60 or greater than 140/90.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harikesh Subramanian, MBBS, Principal Investigator — UPMC Department of Anesthesiology and Perioperative Medicine
Locations (2):
- United States (2):
  - UPMC Montefiore Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perrier ET. Shifting Focus: From Hydration for Performance to Hydration for Health. Ann Nutr Metab. 2017;70 Suppl 1:4-12. doi: 10.1159/000462996. Epub 2017 Jun 15. PMID 28614817
- [Background] Liska D, Mah E, Brisbois T, Barrios PL, Baker LB, Spriet LL. Narrative Review of Hydration and Selected Health Outcomes in the General Population. Nutrients. 2019 Jan 1;11(1):70. doi: 10.3390/nu11010070. PMID 30609670
- [Background] Popkin BM, D'Anci KE, Rosenberg IH. Water, hydration, and health. Nutr Rev. 2010 Aug;68(8):439-58. doi: 10.1111/j.1753-4887.2010.00304.x. PMID 20646222
- [Background] Nuccio RP, Barnes KA, Carter JM, Baker LB. Fluid Balance in Team Sport Athletes and the Effect of Hypohydration on Cognitive, Technical, and Physical Performance. Sports Med. 2017 Oct;47(10):1951-1982. doi: 10.1007/s40279-017-0738-7. PMID 28508338
- [Background] Von Duvillard SP, Braun WA, Markofski M, Beneke R, Leithauser R. Fluids and hydration in prolonged endurance performance. Nutrition. 2004 Jul-Aug;20(7-8):651-6. doi: 10.1016/j.nut.2004.04.011. PMID 15212747
- [Background] American College of Sports Medicine; Sawka MN, Burke LM, Eichner ER, Maughan RJ, Montain SJ, Stachenfeld NS. American College of Sports Medicine position stand. Exercise and fluid replacement. Med Sci Sports Exerc. 2007 Feb;39(2):377-90. doi: 10.1249/mss.0b013e31802ca597. PMID 17277604
- [Background] Lee EC, Fragala MS, Kavouras SA, Queen RM, Pryor JL, Casa DJ. Biomarkers in Sports and Exercise: Tracking Health, Performance, and Recovery in Athletes. J Strength Cond Res. 2017 Oct;31(10):2920-2937. doi: 10.1519/JSC.0000000000002122. PMID 28737585
- [Background] Kenefick RW. Drinking Strategies: Planned Drinking Versus Drinking to Thirst. Sports Med. 2018 Mar;48(Suppl 1):31-37. doi: 10.1007/s40279-017-0844-6. PMID 29368181
- [Background] Love TD, Baker DF, Healey P, Black KE. Measured and perceived indices of fluid balance in professional athletes. The use and impact of hydration assessment strategies. Eur J Sport Sci. 2018 Apr;18(3):349-356. doi: 10.1080/17461391.2017.1418910. Epub 2018 Jan 24. PMID 29364084
- [Background] Maughan RJ, Shirreffs SM. Development of hydration strategies to optimize performance for athletes in high-intensity sports and in sports with repeated intense efforts. Scand J Med Sci Sports. 2010 Oct;20 Suppl 2:59-69. doi: 10.1111/j.1600-0838.2010.01191.x. PMID 20840563
- [Background] Evans GH, James LJ, Shirreffs SM, Maughan RJ. Optimizing the restoration and maintenance of fluid balance after exercise-induced dehydration. J Appl Physiol (1985). 2017 Apr 1;122(4):945-951. doi: 10.1152/japplphysiol.00745.2016. Epub 2017 Jan 26. PMID 28126906
- [Background] Pence J, Bloomer RJ. Impact of Nuun Electrolyte Tablets on Fluid Balance in Active Men and Women. Nutrients. 2020 Oct 2;12(10):3030. doi: 10.3390/nu12103030. PMID 33023276
- [Background] Maughan RJ, Watson P, Cordery PA, Walsh NP, Oliver SJ, Dolci A, Rodriguez-Sanchez N, Galloway SD. A randomized trial to assess the potential of different beverages to affect hydration status: development of a beverage hydration index. Am J Clin Nutr. 2016 Mar;103(3):717-23. doi: 10.3945/ajcn.115.114769. Epub 2015 Dec 23. PMID 26702122

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All enrolled participants completed 3 separate visits in a crossover design, each visit consisting of a different intervention. All participants completed the visits and interventions in the same order as listed below.
Groups:
- Buoy Electrolyte Then Water Only Then Nuun Electrolyte: Visit 1 - Buoy Electrolyte: Buoy intervention amount is 4% of total body weight given in 16 divided doses over 4 hours. The goal is to give 600mg of Na+ over 4 hours while measuring urine output over 6 hours. Therefore, to safely achieve a total dose 600mg Na+ (6-fold increase from single dose) we will use 4 tsps (18 ml) of Buoy diluted in 1 L of water.
  Visit 2 - Water Alone: Water serves as a control. Participants will ingest the same quantity of water (1 L) at a rate of 6.25% of the calculated amount of water every 15 min for 4 hours.
  Visit 3 - Nuun Electrolyte Tablet: Nuun intervention given as 1L bolus and then free water in divided doses for a total of 4% total body weight. The goal is to give a one-time dose of Nuun (600mg Na+) at the start of the trial, diluted in 1L water to be consumed within 30 min (similar to prior published data, Pence 2020).
Period: Visit 1 : Buoy Electrolyte
Arm/Group | Buoy Electrolyte Then Water Only Then Nuun Electrolyte
Started | 30
Completed | 30
Not Completed | 0
Period: Visit 2: Water Only
Arm/Group | Buoy Electrolyte Then Water Only Then Nuun Electrolyte
Started | 30
Completed | 30
Not Completed | 0
Period: Visit 3: Nuun Electrolyte
Arm/Group | Buoy Electrolyte Then Water Only Then Nuun Electrolyte
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Participants: All enrolled participants completed 3 separate visits, each visit consisting of a different intervention. All participants completed the visits and interventions in the same order as listed below.
  Visit 1 - Buoy Electrolyte: Buoy intervention amount is 4% of total body weight given in 16 divided doses over 4 hours. The goal is to give 600mg of Na+ over 4 hours while measuring urine output over 6 hours. The recommended Buoy dosage is ⅓ tsp in 237 ml of water (50mg Na+) multiple times a day (Table 1). Therefore, to safely achieve a total dose 600mg Na+ (6-fold increase from single dose) we will use 4 tsps (18 ml) of Buoy diluted in 1 L of water.
  Visit 2 - Water Alone: Water serves as a control. Participants will ingest the same quantity of water (1 L) at a rate of 6.25% of the calculated amount of water every 15 min for 4 hours.
  Visit 3 - Nuun Electrolyte Tablet: Nuun intervention given as 1L bolus and then free water in divided doses for a total of 4% total body weight. The goal is to give a one-time dose of Nuun (600mg Na+) at the start of the trial, diluted in 1L water to be consumed within 30 min (similar to prior published data, Pence 2020).
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
Body Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 82.6 (16.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Net Fluid Balance
Description: Determined by subtracting the cumulative urine output from the total fluid load consumed
Time Frame: 360 minutes after ingestion
Measure: Mean (Standard Deviation); unit: Liter
Groups:
- Buoy Hydration Drops: Visit 1 consisted of the Buoy Hydration Drops beverage intervention at a dose containing 600mg/Litre of Na+ over 4 hours. All 30 participants completed visit 1.
- Water Alone - Control: Visit 2 consisted of water alone as a control in which each subject ingested 1L of water at a rate of 6/25% of the calculated amount of water every 15 minutes for 4 hours. All 30 participants completed visit 2.
- Nuun Sport Hydration Tabs: Visit 3 consisted of the Nunn Sport Hydration Tabs in which each subject consumed 1L of water with two dissolved tabs, containing 600mg of Na+ over 30 minutes. All 30 participants completed visit 3.
Arm/Group | Buoy Hydration Drops | Water Alone - Control | Nuun Sport Hydration Tabs
Number analyzed (Participants) | 30 | 30 | 30
Liter | 0.28 (0.28) | 0.05 (0.32) | 0.03 (0.20)

2. Primary Outcome: Electrolytes in Urine
Description: Sodium levels will be measured
Time Frame: Urine will be measured during each visit (three total visits that each last 6 hours)
Measure: Mean (Standard Deviation); unit: milliequivalent/L (meq/L)
Arm/Group | Buoy Hydration Drops | Water Alone - Control | Nuun Sport Hydration Tabs
Number analyzed (Participants) | 30 | 30 | 30
milliequivalent/L (meq/L) | 39 (15) | 58 (21) | 48 (47)

3. Primary Outcome: Urine Osmolarity (mOsm/kg)
Description: Osmolarity measures the concentration of solutes in urine. This is a key indicator of how concentrated or diluted the urine is, which directly reflects hydration status and kidney function. This can fluctuate depending on how much water the kidneys are excreting or retaining.
Time Frame: 360 minutes after ingestion
Measure: Mean (Standard Deviation); unit: milliOsm/kilogram (mOsm/kg)
Arm/Group | Buoy Hydration Drops | Water Alone - Control | Nuun Sport Hydration Tabs
Number analyzed (Participants) | 30 | 30 | 30
milliOsm/kilogram (mOsm/kg) | 1928 (544) | 1666 (454) | 1866 (318)

4. Secondary Outcome: Bio Impedance
Description: Bio impedance measured through difference in body fat % pre- and post-urine
Time Frame: 360-minutes after ingestion
Measure: Mean (Standard Deviation); unit: percentage of body fat difference
Arm/Group | Buoy Hydration Drops | Water Alone - Control | Nuun Sport Hydration Tabs
Number analyzed (Participants) | 30 | 30 | 30
percentage of body fat difference | 0.75 (0.62) | 0.64 (0.65) | 0.44 (0.32)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during each visit (total of 3 visits per participant).
Arm/Group | Buoy Hydration Drops | Water Alone - Control | Nuun Sport Hydration Tabs
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT05768789/Prot_SAP_002.pdf
  • Informed Consent Form (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT05768789/ICF_003.pdf